CLINICAL TRIAL: NCT01709318
Title: A Multicenter, Randomized, Partially-blinded, Phase IIb Dose-finding Study on Ovarian Function, Vaginal Bleeding Pattern, and Pharmacokinetics Associated With the Use of Combined Vaginal Rings Releasing 17β-estradiol Plus Three Different Doses of Either Nomegestrol Acetate or Etonogestrel in Healthy Women Aged 18-35 Years. Protocol MK-8175A/MK-8342B 012
Brief Title: A Dose-Finding Study to Evaluate Ovarian Function and Vaginal Bleeding in Next Generation Rings (P06109/MK-8175A/MK-8342B-012)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P06109; 2012-002459-41 (Other: EudraCT Number); P06109 (Other: Schering-Plough); MK-8175A/MK-8342B-012 (Other: Merck)
Record Dates: First submitted 2012-10-16; First posted 2012-10-18 (Estimated); Results first posted 2019-12-05 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2022-02

CONDITIONS: Contraception
MeSH Terms: interventions — nomegestrol acetate; etonogestrel; Ethinyl Estradiol; Estradiol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (7):
- Nomegestrol Acetate-17β-Estradiol (NOMAC-E2) 500/300 μg/day (Experimental): Participants will receive nomegestrol acetate 17β-estradiol (NOMAC-E2) 500/300 μg for three treatment periods, each 28-day treatment period (cycle) consisting of 21 days of vaginal ring use followed by 7 vaginal ring-free days.
  Interventions: Drug: Nomegestrol acetate (NOMAC); Drug: Estradiol (E2)
- Nomegestrol Acetate-17β-Estradiol (NOMAC-E2) 700/300 μg/day (Experimental): Participants will receive nomegestrol acetate 17β-estradiol (NOMAC-E2) 700/300 μg for three treatment periods, each 28-day treatment period (cycle) consisting of 21 days of vaginal ring use followed by 7 vaginal ring-free days.
  Interventions: Drug: Nomegestrol acetate (NOMAC); Drug: Estradiol (E2)
- Nomegestrol Acetate-17β-Estradiol (NOMAC-E2) 900/300 μg/day (Experimental): Participants will receive nomegestrol acetate 17β-estradiol (NOMAC-E2) 900/300 μg for three treatment periods, each 28-day treatment period (cycle) consisting of 21 days of vaginal ring use followed by 7 vaginal ring-free days.
  Interventions: Drug: Nomegestrol acetate (NOMAC); Drug: Estradiol (E2)
- Etonogestrel-17β-Estradiol (ENG-E2) 75/300 μg/day (Experimental): Participants will receive etonogestrel 17β-estradiol (ENG-E2) 75/300 μg for three treatment periods, each 28-day treatment period (cycle) consisting of 21 days of vaginal ring use followed by 7 vaginal ring-free days.
  Interventions: Drug: Etonogestrel (ENG); Drug: Estradiol (E2)
- Etonogestrel-17β-Estradiol (ENG-E2) 100/300 μg/day (Experimental): Participants will receive etonogestrel 17β-estradiol (ENG-E2) 100/300 μg for three treatment periods, each 28-day treatment period (cycle) consisting of 21 days of vaginal ring use followed by 7 vaginal ring-free days.
  Interventions: Drug: Etonogestrel (ENG); Drug: Estradiol (E2)
- Etonogestrel-17β-Estradiol (ENG-E2) 125/300 μg/day (Experimental): Participants will receive etonogestrel 17β-estradiol (ENG-E2)125/300 μg for three 28-day treatment periods, each treatment period (cycle) consisting of 21 days of vaginal ring use followed by 7 vaginal ring-free days.
  Interventions: Drug: Etonogestrel (ENG); Drug: Estradiol (E2)
- NuvaRing® (Active Comparator): Participants will receive NuvaRing® (etonogestrel-ethinyl estradiol [ENG-EE] 120/15 μg) for three treatment periods, each 28-day treatment period (cycle) consisting of 21 days of vaginal ring use followed by 7 vaginal ring-free days.
  Interventions: Drug: Etonogestrel (ENG); Drug: Ethinyl estradiol (EE)

INTERVENTIONS:
Drug: Nomegestrol acetate (NOMAC) — Daily release of 500, 700, or 900 μg.
  Arms: Nomegestrol Acetate-17β-Estradiol (NOMAC-E2) 500/300 μg/day; Nomegestrol Acetate-17β-Estradiol (NOMAC-E2) 700/300 μg/day; Nomegestrol Acetate-17β-Estradiol (NOMAC-E2) 900/300 μg/day
Drug: Etonogestrel (ENG) — Daily release of 75, 100, 120 or 125 μg
  Arms: Etonogestrel-17β-Estradiol (ENG-E2) 100/300 μg/day; Etonogestrel-17β-Estradiol (ENG-E2) 125/300 μg/day; Etonogestrel-17β-Estradiol (ENG-E2) 75/300 μg/day; NuvaRing®
Drug: Ethinyl estradiol (EE) — Daily release of 15 μg
  Arms: NuvaRing®
Drug: Estradiol (E2) — Daily release of 300 μg
  Arms: Etonogestrel-17β-Estradiol (ENG-E2) 100/300 μg/day; Etonogestrel-17β-Estradiol (ENG-E2) 125/300 μg/day; Etonogestrel-17β-Estradiol (ENG-E2) 75/300 μg/day; Nomegestrol Acetate-17β-Estradiol (NOMAC-E2) 500/300 μg/day; Nomegestrol Acetate-17β-Estradiol (NOMAC-E2) 700/300 μg/day; Nomegestrol Acetate-17β-Estradiol (NOMAC-E2) 900/300 μg/day

SUMMARY:
The primary objective of this trial was to identify at least one next generation ring (NGR) that demonstrates inhibition of ovulation (which was considered confirmed if in the subset of participants ovulation was observed in less than 15% of the participants at any time during the 3 treatment cycles of the study) and cycle control that was non-inferior to NuvaRing®, as judged by the incidence of breakthrough bleeding and/or spotting (BTB-S) during Cycle 3. The primary hypothesis was that at least 1 of the 6 NGRs would show inhibition of ovulation and cycle control during Treatment Cycle 3 that is non-inferior to NuvaRing®, as judged by the incidence of BTB-S.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) ≥18 and ≤35
* Regular cycles from 24 to 35 days in length, with an intra-individual variation of ±3 days permitted within this range
* Good physical and mental health

Exclusion Criteria:

* Diabetes mellitus with vascular involvement
* Presence of a severe or multiple risk factor(s) for venous or arterial thrombosis
* Severe dyslipoproteinemia
* Severe hypertension
* Presence or history of pancreatitis associated with severe hypertriglyceridaemia
* Presence or history of severe hepatic disease
* Undiagnosed vaginal bleeding
* Known or suspected pregnancy
* Participation in another investigational drug study within 30 days prior to screening visit
* History of malignancy ≤5 years, except for adequately treated basal cell or squamous cell skin cancer, or in situ cervical cancer
* Documented abnormal cervical smear result in 6 months prior to screening visit
* Sterilization using a fallopian tube occlusion device (e.g., Essure method)
* Sex hormone therapy within 2 months prior to screening visit for purpose other than contraception, or injectable hormonal contraception within 6 months prior to screening

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 666 (Actual)
Dates: Start 2012-12-12 (Actual); Primary Completion 2013-10-22 (Actual); Study Completion 2013-10-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Duijkers I, Klipping C, Heger-Mahn D, Fayad GN, Frenkl TL, Cruz SM, Korver T. Phase II dose-finding study on ovulation inhibition and cycle control associated with the use of contraceptive vaginal rings containing 17beta-estradiol and the progestagens etonogestrel or nomegestrol acetate compared to NuvaRing. Eur J Contracept Reprod Health Care. 2018 Aug;23(4):245-254. doi: 10.1080/13625187.2018.1506101. Epub 2018 Sep 11. PMID 30203681

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study enrolled healthy female participants aged 18 to 35 years, with cycles between 24 to 35 days in length.
Pre-assignment Details: Of the 757 participants who were screened for inclusion in the trial, 666 participants were randomized, and 660 participants were treated.
Groups:
- Nomegestrol Acetate-17β-Estradiol (NOMAC-E2) 500/300 μg/Day: Participants received nomegestrol acetate-17β-estradiol (NOMAC-E2) 500/300 μg for three treatment periods, each 28-day treatment period (cycle) consisting of 21 days of vaginal ring use followed by 7 vaginal ring-free days.
- Nomegestrol Acetate-17β-Estradiol (NOMAC-E2) 700/300 μg/Day: Participants received nomegestrol acetate-17β-estradiol (NOMAC-E2) 700/300 μg for three treatment periods, each 28-day treatment period (cycle) consisting of 21 days of vaginal ring use followed by 7 vaginal ring-free days.
- Nomegestrol Acetate-17β-Estradiol (NOMAC-E2) 900/300 μg/Day: Participants received nomegestrol acetate-17β-estradiol (NOMAC-E2) 900/300 μg for three treatment periods, each 28-day treatment period (cycle) consisting of 21 days of vaginal ring use followed by 7 vaginal ring-free days.
- Etonogestrel-17β-Estradiol (ENG-E2) 75/300 μg/Day: Participants received etonogestrel-17β-estradiol (ENG-E2) 75/300 μg for three treatment periods, each 28-day treatment period (cycle) consisting of 21 days of vaginal ring use followed by 7 vaginal ring-free days.
- Etonogestrel-17β-Estradiol (ENG-E2) 100/300 μg/Day: Participants received etonogestrel-17β-estradiol (ENG-E2) 100/300 μg for three treatment periods, each 28-day treatment period (cycle) consisting of 21 days of vaginal ring use followed by 7 vaginal ring-free days.
- Etonogestrel-17β-Estradiol (ENG-E2) 125/300 μg/Day: Participants received etonogestrel-17β-estradiol (ENG-E2) 125/300 μg for three 28-day treatment periods, each treatment period (cycle) consisting of 21 days of vaginal ring use followed by 7 vaginal ring-free days.
- NuvaRing®: Participants received NuvaRing® (etonogestrel-ethinyl estradiol [ENG-EE] 120/15 μg) for three treatment periods, each 28-day treatment period (cycle) consisting of 21 days of vaginal ring use followed by 7 vaginal ring-free days.
Period: Overall Study
Arm/Group | Nomegestrol Acetate-17β-Estradiol (NOMAC-E2) 500/300 μg/Day | Nomegestrol Acetate-17β-Estradiol (NOMAC-E2) 700/300 μg/Day | Nomegestrol Acetate-17β-Estradiol (NOMAC-E2) 900/300 μg/Day | Etonogestrel-17β-Estradiol (ENG-E2) 75/300 μg/Day | Etonogestrel-17β-Estradiol (ENG-E2) 100/300 μg/Day | Etonogestrel-17β-Estradiol (ENG-E2) 125/300 μg/Day | NuvaRing®
Started | 82 | 85 | 77 | 78 | 78 | 84 | 182
Treated | 79 | 85 | 78 | 77 | 77 | 86 | 178
Completed | 73 | 78 | 71 | 72 | 74 | 80 | 171
Not Completed | 9 | 7 | 6 | 6 | 4 | 4 | 11
Not completed — Adverse Event | 3 | 4 | 2 | 2 | 0 | 1 | 2
Not completed — Lost to Follow-up | 2 | 0 | 0 | 0 | 1 | 1 | 1
Not completed — Non-compliance with Study Drug | 0 | 2 | 1 | 1 | 0 | 0 | 2
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Pregnancy | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 2 | 0 | 1
Not completed — Technical Problems | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 0 | 3 | 3 | 0 | 2 | 4
Not completed — Other Protocol Specified Criteria | 0 | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: 4 participants used the incorrect vaginal ring per the randomization schedule throughout the trial (2 participants in ENG-E2 125/300 μg and 1 participant each in the NOMAC-E2 900/300 μg and NuvaRing group).
Groups:
- Total: Total of all reporting groups
Arm/Group | Nomegestrol Acetate-17β-Estradiol (NOMAC-E2) 500/300 μg/Day | Nomegestrol Acetate-17β-Estradiol (NOMAC-E2) 700/300 μg/Day | Nomegestrol Acetate-17β-Estradiol (NOMAC-E2) 900/300 μg/Day | Etonogestrel-17β-Estradiol (ENG-E2) 75/300 μg/Day | Etonogestrel-17β-Estradiol (ENG-E2) 100/300 μg/Day | Etonogestrel-17β-Estradiol (ENG-E2) 125/300 μg/Day | NuvaRing® | Total
Number analyzed (Participants) | 79 | 85 | 78 | 77 | 77 | 86 | 178 | 660
Age, Continuous [Mean (Standard Deviation); unit: Years] | 26.7 (5.02) | 26.7 (4.91) | 26.1 (4.46) | 25.5 (4.87) | 26.1 (4.52) | 27.1 (4.61) | 25.9 (4.82) | 26.3 (4.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 79 | 85 | 78 | 77 | 77 | 86 | 178 | 660
  Male | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Black or African American | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 4
  White | 77 | 83 | 76 | 73 | 77 | 85 | 174 | 645
  More than one race | 1 | 0 | 2 | 2 | 0 | 1 | 2 | 8
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Ovulation Incidence, by Cycle
Description: Ovulation was defined as having 2 or more consecutive progesterone concentrations >16 nmol/L within 5 days, confirmed by ultrasound evidence of ovulation (follicular rupture or preceding presence of a follicle-like structure >15 mm in size).
Time Frame: Day 1 of Treatment Cycle 1 through Day 28 of Treatment Cycle 3 (Up to ~92 days)
Population: The analysis population included all participants in whom vaginal rings were inserted and received ultrasound and hormonal assessments, excluding participants who were protocol violators in terms of ring use, daily diary entry or prohibited medications.
Measure: Number; unit: Percentage of Participants
Arm/Group | Nomegestrol Acetate-17β-Estradiol (NOMAC-E2) 500/300 μg/Day | Nomegestrol Acetate-17β-Estradiol (NOMAC-E2) 700/300 μg/Day | Nomegestrol Acetate-17β-Estradiol (NOMAC-E2) 900/300 μg/Day | Etonogestrel-17β-Estradiol (ENG-E2) 75/300 μg/Day | Etonogestrel-17β-Estradiol (ENG-E2) 100/300 μg/Day | Etonogestrel-17β-Estradiol (ENG-E2) 125/300 μg/Day | NuvaRing®
Number analyzed (Participants) | 65 | 73 | 57 | 60 | 63 | 65 | 126
Percentage of Participants
  Cycle 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Cycle 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Cycle 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Percentage of Participants With Progesterone Concentrations >16 Nmol/L, by Cycle
Description: Maximum progesterone (Max P) was defined as the maximum progesterone value. Ovulation was defined as 2 or more consecutive progesterone concentrations >16 nmol/L within 5 days during the 3 treatment cycles, supported by ultrasound evidence of ovulation. The Max P values greater than 16 nmol/L are presented by vaginal ring group and cycle.
Time Frame: Day 1 of Treatment Cycle 1 through Day 28 of Treatment Cycle 3 (Up to ~92 days)
Population: The analysis population included all participants in whom vaginal rings were inserted and received hormonal assessment for progesterone concentration, excluding participants who were protocol violators in terms of ring use, daily diary entry or prohibited medications.
Measure: Number; unit: Percentage of Participants
Arm/Group | Nomegestrol Acetate-17β-Estradiol (NOMAC-E2) 500/300 μg/Day | Nomegestrol Acetate-17β-Estradiol (NOMAC-E2) 700/300 μg/Day | Nomegestrol Acetate-17β-Estradiol (NOMAC-E2) 900/300 μg/Day | Etonogestrel-17β-Estradiol (ENG-E2) 75/300 μg/Day | Etonogestrel-17β-Estradiol (ENG-E2) 100/300 μg/Day | Etonogestrel-17β-Estradiol (ENG-E2) 125/300 μg/Day | NuvaRing®
Number analyzed (Participants) | 65 | 73 | 57 | 60 | 63 | 65 | 126
Percentage of Participants
  Cycle 1 Max P > 16 nmol/L: number analyzed (Participants) | 18 | 19 | 19 | 20 | 19 | 19 | 21
  Cycle 1 Max P > 16 nmol/L | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Cycle 2 Max P > 16 nmol/L: number analyzed (Participants) | 17 | 16 | 16 | 20 | 19 | 17 | 19
  Cycle 2 Max P > 16 nmol/L | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Cycle 3 Max P > 16 nmol/L: number analyzed (Participants) | 17 | 15 | 14 | 17 | 19 | 17 | 19
  Cycle 3 Max P > 16 nmol/L | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Percentage of Participants With Breakthrough Bleeding and/or Spotting During Cycle 3
Description: Breakthrough bleeding and/or spotting (BTB-S) is defined as any bleeding or spotting episode that occurred during the expected non-bleeding period that was neither an early nor a continued withdrawal bleeding. Bleeding = any bloody vaginal discharge that required one or more sanitary pads or tampons per day; Spotting = any bloody vaginal discharge that required no sanitary pads or tampons per day.
Time Frame: Day 1 Cycle 3 through Day 28 Cycle 3 (Up to ~28 days)
Population: The analysis population included all participants in whom vaginal rings were inserted and had an evaluable cycle with non-missing bleeding data in the respective cycle, excluding participants who were protocol violators in terms of ring use, daily diary entry or prohibited medications.
Measure: Number; unit: Percentage of Participants
Arm/Group | Nomegestrol Acetate-17β-Estradiol (NOMAC-E2) 500/300 μg/Day | Nomegestrol Acetate-17β-Estradiol (NOMAC-E2) 700/300 μg/Day | Nomegestrol Acetate-17β-Estradiol (NOMAC-E2) 900/300 μg/Day | Etonogestrel-17β-Estradiol (ENG-E2) 75/300 μg/Day | Etonogestrel-17β-Estradiol (ENG-E2) 100/300 μg/Day | Etonogestrel-17β-Estradiol (ENG-E2) 125/300 μg/Day | NuvaRing®
Number analyzed (Participants) | 48 | 45 | 40 | 44 | 49 | 47 | 97
Percentage of Participants | 14.6 | 13.3 | 17.5 | 13.6 | 16.3 | 6.4 | 6.2
Statistical Analysis 1: Comparison: Nomegestrol Acetate-17β-Estradiol (NOMAC-E2) 500/300 μg/Day vs NuvaRing®; Test type: Non-Inferiority — Based on a longitudinal data analysis (LDA) model with terms for treatment, cycle and the interaction cycle by treatment and stratum:starter/switcher followed by Miettinen and Nurminen's method. Non-inferiority criterion was met if the upper bound of the 95% CI of the difference is less than or equal to 10%; Difference in Percent = 8.3, 95% CI 2-sided [-4.3 to 26.5] — 95% CI adjusted for multiplicity (Dunnett)
Statistical Analysis 2: Comparison: Nomegestrol Acetate-17β-Estradiol (NOMAC-E2) 700/300 μg/Day vs NuvaRing®; Test type: Non-Inferiority — Based on a LDA model with terms for treatment, cycle and the interaction cycle by treatment and stratum:starter/switcher followed by Miettinen and Nurminen's method. Non-inferiority criterion was met if the upper bound of the 95% CI of the difference is less than or equal to 10%; Difference in Percent = 6.5, 95% CI 2-sided [-5.7 to 24.8] — 95% CI adjusted for multiplicity (Dunnett)
Statistical Analysis 3: Comparison: Nomegestrol Acetate-17β-Estradiol (NOMAC-E2) 900/300 μg/Day vs NuvaRing®; Test type: Non-Inferiority — [test comment as in outcome 3, analysis 2]; Difference in Percent = 12.3, 95% CI 2-sided [-1.7 to 33.1] — 95% CI adjusted for multiplicity (Dunnett)
Statistical Analysis 4: Comparison: Etonogestrel-17β-Estradiol (ENG-E2) 75/300 μg/Day vs NuvaRing®; Test type: Non-Inferiority — [test comment as in outcome 3, analysis 2]; Difference in Percent = 6.6, 95% CI 2-sided [-5.7 to 25.4] — 95% CI adjusted for multiplicity (Dunnett)
Statistical Analysis 5: Comparison: Etonogestrel-17β-Estradiol (ENG-E2) 100/300 μg/Day vs NuvaRing®; Test type: Non-Inferiority — [test comment as in outcome 3, analysis 2]; Difference in Percent = 9.3, 95% CI 2-sided [-3.5 to 27.4] — 95% CI adjusted for multiplicity (Dunnett)
Statistical Analysis 6: Comparison: Etonogestrel-17β-Estradiol (ENG-E2) 125/300 μg/Day vs NuvaRing®; Test type: Non-Inferiority — [test comment as in outcome 3, analysis 2]; Difference in Percent = -0.0, 95% CI 2-sided [-10.7 to 15.9] — 95% CI adjusted for multiplicity (Dunnett)

4. Secondary Outcome: Percentage of Participants With Absence of Withdrawal Bleeding and/or Spotting During Cycle 2
Description: Withdrawal bleeding and/or spotting is considered any bleeding or spotting episode that starts during or continues into the expected bleeding period (i.e., when the ring has been removed the last week of the cycle). Absence of withdrawal bleeding is no withdrawal bleeding and/or spotting episodes during an expected bleeding period when the ring has been removed.
Time Frame: Day 1 Cycle 2 through Day 28 Cycle 2 (Up to ~28 days)
Population: as for outcome 3
Measure: Number; unit: Percentage of Participants
Arm/Group | Nomegestrol Acetate-17β-Estradiol (NOMAC-E2) 500/300 μg/Day | Nomegestrol Acetate-17β-Estradiol (NOMAC-E2) 700/300 μg/Day | Nomegestrol Acetate-17β-Estradiol (NOMAC-E2) 900/300 μg/Day | Etonogestrel-17β-Estradiol (ENG-E2) 75/300 μg/Day | Etonogestrel-17β-Estradiol (ENG-E2) 100/300 μg/Day | Etonogestrel-17β-Estradiol (ENG-E2) 125/300 μg/Day | NuvaRing®
Number analyzed (Participants) | 55 | 53 | 45 | 51 | 54 | 52 | 111
Percentage of Participants | 5.5 | 1.9 | 4.4 | 7.8 | 3.7 | 1.9 | 1.8
Statistical Analysis 1: Comparison: Nomegestrol Acetate-17β-Estradiol (NOMAC-E2) 500/300 μg/Day vs NuvaRing®; Test type: Non-Inferiority — [test comment as in outcome 3, analysis 2]; Difference in Percent = 3.2, 95% CI 2-sided [-3.6 to 16.4] — 95% CI adjusted for multiplicity (Dunnett)
Statistical Analysis 2: Comparison: Nomegestrol Acetate-17β-Estradiol (NOMAC-E2) 700/300 μg/Day vs NuvaRing®; Test type: Non-Inferiority — [test comment as in outcome 3, analysis 2]; Difference in Percent = -0.0, 95% CI 2-sided [-6.2 to 11.0] — 95% CI adjusted for multiplicity (Dunnett)
Statistical Analysis 3: Comparison: Nomegestrol Acetate-17β-Estradiol (NOMAC-E2) 900/300 μg/Day vs NuvaRing®; Test type: Non-Inferiority — [test comment as in outcome 3, analysis 2]; Difference in Percent = 3.0, 95% CI 2-sided [-3.8 to 17.5] — 95% CI adjusted for multiplicity (Dunnett)
Statistical Analysis 4: Comparison: Etonogestrel-17β-Estradiol (ENG-E2) 75/300 μg/Day vs NuvaRing®; Test type: Non-Inferiority — [test comment as in outcome 3, analysis 2]; Difference in Percent = 4.7, 95% CI 2-sided [-2.5 to 18.9] — 95% CI adjusted for multiplicity (Dunnett)
Statistical Analysis 5: Comparison: Etonogestrel-17β-Estradiol (ENG-E2) 100/300 μg/Day vs NuvaRing®; Test type: Non-Inferiority — [test comment as in outcome 3, analysis 2]; Difference in Percent = 1.4, 95% CI 2-sided [-5.0 to 13.4] — 95% CI adjusted for multiplicity (Dunnett)
Statistical Analysis 6: Comparison: Etonogestrel-17β-Estradiol (ENG-E2) 125/300 μg/Day vs NuvaRing®; Test type: Non-Inferiority — [test comment as in outcome 3, analysis 2]; Difference in Percent = -0.0, 95% CI 2-sided [-6.2 to 11.0] — 95% CI adjusted for multiplicity (Dunnett)

5. Secondary Outcome: Intensity of Withdrawal Bleeding During Cycle 2
Description: Intensity of withdrawal bleeding during Cycle 2 was defined as the ratio of the number of withdrawal bleeding days divided by the number of withdrawal bleeding and/or spotting days. Withdrawal bleeding and/or spotting is considered any bleeding or spotting episode that starts during or continues into the expected bleeding period (i.e., when the ring has been removed the last week of the cycle). Absence of withdrawal bleeding is no withdrawal bleeding and/or spotting episodes during an expected bleeding period when the ring has been removed.
Time Frame: Day 1 Cycle 2 through Day 28 Cycle 2 (Up to ~28 days)
Population: The analysis population included all participants in whom vaginal rings were inserted and had an evaluable cycle with non-missing bleeding data in the respective cycle, and with at least one withdrawal bleeding or spotting day, excluding participants who were protocol violators in terms of ring use, daily diary entry or prohibited medications.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Nomegestrol Acetate-17β-Estradiol (NOMAC-E2) 500/300 μg/Day | Nomegestrol Acetate-17β-Estradiol (NOMAC-E2) 700/300 μg/Day | Nomegestrol Acetate-17β-Estradiol (NOMAC-E2) 900/300 μg/Day | Etonogestrel-17β-Estradiol (ENG-E2) 75/300 μg/Day | Etonogestrel-17β-Estradiol (ENG-E2) 100/300 μg/Day | Etonogestrel-17β-Estradiol (ENG-E2) 125/300 μg/Day | NuvaRing®
Number analyzed (Participants) | 52 | 52 | 43 | 47 | 52 | 51 | 109
Ratio | 0.87 (0.25) | 0.92 (0.17) | 0.86 (0.19) | 0.90 (0.18) | 0.92 (0.18) | 0.93 (0.14) | 0.95 (0.12)
Statistical Analysis 1: Comparison: Nomegestrol Acetate-17β-Estradiol (NOMAC-E2) 500/300 μg/Day vs NuvaRing®; Test type: Other — Based on longitudinal data analysis (LDA) model: generalized linear mixed model with terms for stratum, ring group, cycle (and the interaction of cycle by ring group), and continuous response variable; p = 0.096, LDA; Difference of Least Squares (LS) Mean = -0.08
Statistical Analysis 2: Comparison: Nomegestrol Acetate-17β-Estradiol (NOMAC-E2) 700/300 μg/Day vs NuvaRing®; Test type: Other — Based on longitudinal data analysis model: generalized linear mixed model with terms for stratum, ring group, cycle (and the interaction of cycle by ring group), and continuous response variable; p = 0.993, LDA; Difference of LS Mean = -0.03
Statistical Analysis 3: Comparison: Nomegestrol Acetate-17β-Estradiol (NOMAC-E2) 900/300 μg/Day vs NuvaRing®; Test type: Other — [test comment as in outcome 5, analysis 2]; p = 0.124, LDA; Difference of LS Mean = -0.08
Statistical Analysis 4: Comparison: Etonogestrel-17β-Estradiol (ENG-E2) 75/300 μg/Day vs NuvaRing®; Test type: Other — [test comment as in outcome 5, analysis 2]; p = 0.845, LDA; Difference of LS Mean = -0.05
Statistical Analysis 5: Comparison: Etonogestrel-17β-Estradiol (ENG-E2) 100/300 μg/Day vs NuvaRing®; Test type: Other — [test comment as in outcome 5, analysis 2]; p = 0.976, LDA; Difference of LS Mean = -0.04
Statistical Analysis 6: Comparison: Etonogestrel-17β-Estradiol (ENG-E2) 125/300 μg/Day vs NuvaRing®; Test type: Other — [test comment as in outcome 5, analysis 2]; p = 0.995, LDA; Difference of LS Mean = -0.03

6. Secondary Outcome: Intensity of Breakthrough Bleeding and/or Spotting During Cycle 3
Description: Intensity of breakthrough bleeding and/or spotting (BTB-S) during Cycle 3 was defined as the ratio of the number of breakthrough bleeding days divided by the number of breakthrough bleeding and/or spotting days. Breakthrough bleeding and/or spotting (BTB-S) is defined as any bleeding or spotting episode that occurred during the expected non-bleeding period that was neither an early nor a continued withdrawal bleeding. Bleeding = any bloody vaginal discharge that required one or more sanitary pads or tampons per day; Spotting = any bloody vaginal discharge that required no sanitary pads or tampons per day.
Time Frame: Day 1 Cycle 3 through Day 28 Cycle 3 (Up to ~ 28 days)
Population: The analysis population included all participants in whom vaginal rings were inserted and had an evaluable cycle with non-missing bleeding data in the respective cycle, and with at least one breakthrough bleeding and/or spotting day, excluding protocol violators in terms of ring use, daily diary entry or prohibited medications.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Nomegestrol Acetate-17β-Estradiol (NOMAC-E2) 500/300 μg/Day | Nomegestrol Acetate-17β-Estradiol (NOMAC-E2) 700/300 μg/Day | Nomegestrol Acetate-17β-Estradiol (NOMAC-E2) 900/300 μg/Day | Etonogestrel-17β-Estradiol (ENG-E2) 75/300 μg/Day | Etonogestrel-17β-Estradiol (ENG-E2) 100/300 μg/Day | Etonogestrel-17β-Estradiol (ENG-E2) 125/300 μg/Day | NuvaRing®
Number analyzed (Participants) | 7 | 6 | 7 | 6 | 8 | 3 | 6
Ratio | 0.42 (0.45) | 0.80 (0.40) | 0.68 (0.47) | 0.73 (0.16) | 0.67 (0.43) | 0.33 (0.58) | 0.67 (0.52)
Statistical Analysis 1: Comparison: Nomegestrol Acetate-17β-Estradiol (NOMAC-E2) 500/300 μg/Day vs NuvaRing®; Test type: Other — [test comment as in outcome 5, analysis 1]; p = 1.000, LDA; Difference of Least Squares (LS) Mean = -0.01
Statistical Analysis 2: Comparison: Nomegestrol Acetate-17β-Estradiol (NOMAC-E2) 700/300 μg/Day vs NuvaRing®; Test type: Other — [test comment as in outcome 5, analysis 2]; p = 0.996, LDA; Difference of LS Mean = 0.19
Statistical Analysis 3: Comparison: Nomegestrol Acetate-17β-Estradiol (NOMAC-E2) 900/300 μg/Day vs NuvaRing®; Test type: Other — [test comment as in outcome 5, analysis 2]; p = 1.000, LDA; Difference of LS Mean = -0.06
Statistical Analysis 4: Comparison: Etonogestrel-17β-Estradiol (ENG-E2) 75/300 μg/Day vs NuvaRing®; Test type: Other — [test comment as in outcome 5, analysis 2]; p = 1.000, LDA; Difference of LS Mean = -0.04
Statistical Analysis 5: Comparison: Etonogestrel-17β-Estradiol (ENG-E2) 100/300 μg/Day vs NuvaRing®; Test type: Other — [test comment as in outcome 5, analysis 2]; p = 1.000, LDA; Difference of LS Mean = 0.09
Statistical Analysis 6: Comparison: Etonogestrel-17β-Estradiol (ENG-E2) 125/300 μg/Day vs NuvaRing®; Test type: Other — [test comment as in outcome 5, analysis 2]; p = 0.998, LDA; Difference of LS Mean = -0.24

7. Other Pre Specified Outcome: Number of Participants With Venous or Arterial Thrombotic/Thromboembolic Events
Description: Venous or arterial thrombotic/thrombo-embolic events, (VTEs or ATEs) (e.g., deep venous thrombosis, pulmonary embolism, myocardial infarction, cerebrovascular accident) were assessed.
Time Frame: From Cycle 1 Day 1 up to 8 days after Day 28 of Cycle 3 (Up to ~92 days)
Population: The analysis population included all randomized participants in whom a vaginal ring was inserted.
Measure: Count of Participants; unit: Participants
Arm/Group | Nomegestrol Acetate-17β-Estradiol (NOMAC-E2) 500/300 μg/Day | Nomegestrol Acetate-17β-Estradiol (NOMAC-E2) 700/300 μg/Day | Nomegestrol Acetate-17β-Estradiol (NOMAC-E2) 900/300 μg/Day | Etonogestrel-17β-Estradiol (ENG-E2) 75/300 μg/Day | Etonogestrel-17β-Estradiol (ENG-E2) 100/300 μg/Day | Etonogestrel-17β-Estradiol (ENG-E2) 125/300 μg/Day | NuvaRing®
Number analyzed (Participants) | 79 | 85 | 78 | 77 | 77 | 86 | 178
Participants | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0

8. Secondary Outcome: Percentage of Participants Who Experienced At Least One Adverse Event
Description: An adverse event (AE) is defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a study drug, whether or not it is considered related to the study drug.
Time Frame: Up to ~92 days
Population: The analysis population included all randomized participants in whom a vaginal ring was inserted.
Measure: Number; unit: Percentage of Participants
Arm/Group | Nomegestrol Acetate-17β-Estradiol (NOMAC-E2) 500/300 μg/Day | Nomegestrol Acetate-17β-Estradiol (NOMAC-E2) 700/300 μg/Day | Nomegestrol Acetate-17β-Estradiol (NOMAC-E2) 900/300 μg/Day | Etonogestrel-17β-Estradiol (ENG-E2) 75/300 μg/Day | Etonogestrel-17β-Estradiol (ENG-E2) 100/300 μg/Day | Etonogestrel-17β-Estradiol (ENG-E2) 125/300 μg/Day | NuvaRing®
Number analyzed (Participants) | 79 | 85 | 78 | 77 | 77 | 86 | 178
Percentage of Participants | 43.0 | 40.0 | 43.6 | 37.7 | 39.0 | 46.5 | 39.3

9. Secondary Outcome: Percentage of Participants Who Experienced At Least One Serious Adverse Event
Description: A serious adverse event (SAE) is an AE that results in death, is life threatening, requires or prolongs an existing hospitalization, results in persistent or significant disability or incapacity, is a congenital anomaly or birth defect, is a cancer, is associated with an overdose; or is another important medical event deemed such by medical or scientific judgment.
Time Frame: Up to ~92 days
Population: The analysis population included all randomized participants in whom a vaginal ring was inserted.
Measure: Number; unit: Percentage of Participants
Arm/Group | Nomegestrol Acetate-17β-Estradiol (NOMAC-E2) 500/300 μg/Day | Nomegestrol Acetate-17β-Estradiol (NOMAC-E2) 700/300 μg/Day | Nomegestrol Acetate-17β-Estradiol (NOMAC-E2) 900/300 μg/Day | Etonogestrel-17β-Estradiol (ENG-E2) 75/300 μg/Day | Etonogestrel-17β-Estradiol (ENG-E2) 100/300 μg/Day | Etonogestrel-17β-Estradiol (ENG-E2) 125/300 μg/Day | NuvaRing®
Number analyzed (Participants) | 79 | 85 | 78 | 77 | 77 | 86 | 178
Percentage of Participants | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0

10. Secondary Outcome: Percentage of Participants Who Experienced At Least One Drug-Related Adverse Event
Description: An adverse event (AE) is defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a study drug, whether or not it is considered related to the study drug. A drug-related AE was defined as any AE for which there is reasonable possibility of drug relationship as assessed by the Investigator.
Time Frame: Up to ~92 days
Population: The analysis population included all randomized participants in whom a vaginal ring was inserted.
Measure: Number; unit: Percentage of Participants
Arm/Group | Nomegestrol Acetate-17β-Estradiol (NOMAC-E2) 500/300 μg/Day | Nomegestrol Acetate-17β-Estradiol (NOMAC-E2) 700/300 μg/Day | Nomegestrol Acetate-17β-Estradiol (NOMAC-E2) 900/300 μg/Day | Etonogestrel-17β-Estradiol (ENG-E2) 75/300 μg/Day | Etonogestrel-17β-Estradiol (ENG-E2) 100/300 μg/Day | Etonogestrel-17β-Estradiol (ENG-E2) 125/300 μg/Day | NuvaRing®
Number analyzed (Participants) | 79 | 85 | 78 | 77 | 77 | 86 | 178
Percentage of Participants | 26.6 | 23.5 | 26.9 | 29.9 | 26.0 | 31.4 | 20.8

11. Secondary Outcome: Percentage of Participants With Any Drug-Related Serious Adverse Event
Description: A serious adverse event (SAE) is an AE that results in death, is life threatening, requires or prolongs an existing hospitalization, results in persistent or significant disability or incapacity, is a congenital anomaly or birth defect, is a cancer, is associated with an overdose; or is another important medical event deemed such by medical or scientific judgment. A drug-related SAE was defined as any SAE for which there is reasonable possibility of drug relationship as assessed by the Investigator.
Time Frame: Up to ~92 days
Population: The analysis population included all randomized participants in whom a vaginal ring was inserted.
Measure: Number; unit: Percentage of Participants
Arm/Group | Nomegestrol Acetate-17β-Estradiol (NOMAC-E2) 500/300 μg/Day | Nomegestrol Acetate-17β-Estradiol (NOMAC-E2) 700/300 μg/Day | Nomegestrol Acetate-17β-Estradiol (NOMAC-E2) 900/300 μg/Day | Etonogestrel-17β-Estradiol (ENG-E2) 75/300 μg/Day | Etonogestrel-17β-Estradiol (ENG-E2) 100/300 μg/Day | Etonogestrel-17β-Estradiol (ENG-E2) 125/300 μg/Day | NuvaRing®
Number analyzed (Participants) | 79 | 85 | 78 | 77 | 77 | 86 | 178
Percentage of Participants | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0

12. Secondary Outcome: Percentage of Participants Who Discontinued Study Drug Due to an Adverse Event
Description: as for outcome 8
Time Frame: Up to ~92 days
Population: The analysis population included all randomized participants in whom a vaginal ring was inserted.
Measure: Number; unit: Percentage of Participants
Arm/Group | Nomegestrol Acetate-17β-Estradiol (NOMAC-E2) 500/300 μg/Day | Nomegestrol Acetate-17β-Estradiol (NOMAC-E2) 700/300 μg/Day | Nomegestrol Acetate-17β-Estradiol (NOMAC-E2) 900/300 μg/Day | Etonogestrel-17β-Estradiol (ENG-E2) 75/300 μg/Day | Etonogestrel-17β-Estradiol (ENG-E2) 100/300 μg/Day | Etonogestrel-17β-Estradiol (ENG-E2) 125/300 μg/Day | NuvaRing®
Number analyzed (Participants) | 79 | 85 | 78 | 77 | 77 | 86 | 178
Percentage of Participants | 3.8 | 4.7 | 2.6 | 2.6 | 0 | 1.2 | 1.1

ADVERSE EVENTS:
Time Frame: Up to ~92 days
Description: The analysis population consisted of all randomized participants in whom a vaginal ring was inserted.
Arm/Group | Nomegestrol Acetate-17β-Estradiol (NOMAC-E2) 500/300 μg/Day | Nomegestrol Acetate-17β-Estradiol (NOMAC-E2) 700/300 μg/Day | Nomegestrol Acetate-17β-Estradiol (NOMAC-E2) 900/300 μg/Day | Etonogestrel-17β-Estradiol (ENG-E2) 75/300 μg/Day | Etonogestrel-17β-Estradiol (ENG-E2) 100/300 μg/Day | Etonogestrel-17β-Estradiol (ENG-E2) 125/300 μg/Day | NuvaRing®
All-Cause Mortality (participants affected / at risk) | 0/79 | 0/85 | 0/78 | 0/77 | 0/77 | 0/86 | 0/178
Serious Adverse Events (participants affected / at risk) | 0/79 | 0/85 | 0/78 | 0/77 | 0/77 | 0/86 | 0/178
Other Adverse Events (participants affected / at risk) | 23/79 | 20/85 | 26/78 | 24/77 | 22/77 | 25/86 | 46/178
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nomegestrol Acetate-17β-Estradiol (NOMAC-E2) 500/300 μg/Day (N=79) | Nomegestrol Acetate-17β-Estradiol (NOMAC-E2) 700/300 μg/Day (N=85) | Nomegestrol Acetate-17β-Estradiol (NOMAC-E2) 900/300 μg/Day (N=78) | Etonogestrel-17β-Estradiol (ENG-E2) 75/300 μg/Day (N=77) | Etonogestrel-17β-Estradiol (ENG-E2) 100/300 μg/Day (N=77) | Etonogestrel-17β-Estradiol (ENG-E2) 125/300 μg/Day (N=86) | NuvaRing® (N=178)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (2) | 6 (9) | 1 (1) | 3 (3) | 2 (3)
Nausea (Gastrointestinal disorders) | 4 (7) | 1 (1) | 2 (2) | 4 (4) | 1 (1) | 1 (1) | 7 (8)
Nasopharyngitis (Infections and infestations) | 9 (12) | 5 (5) | 11 (13) | 11 (14) | 7 (7) | 8 (9) | 16 (18)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0) | 1 (1) | 1 (2) | 2 (3) | 2 (3) | 4 (8)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 12 (24) | 11 (21) | 14 (43) | 13 (35) | 15 (29) | 13 (35) | 24 (47)
Dysmenorrhoea (Reproductive system and breast disorders) | 4 (5) | 2 (2) | 5 (5) | 2 (2) | 3 (3) | 6 (8) | 7 (11)
Vaginal discharge (Reproductive system and breast disorders) | 1 (1) | 6 (9) | 4 (5) | 4 (4) | 5 (9) | 4 (6) | 3 (4)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 1 (2) | 2 (2) | 4 (5) | 1 (1) | 2 (2) | 4 (4)
Acne (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (4) | 6 (8) | 3 (3) | 2 (2) | 6 (10) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines.